CLINICAL TRIAL: NCT06451159
Title: Phase 1, Open-Label, Single Center Study of KYV-101, an Autologous Fully-Human Anti-CD19 Chimeric Antigen Receptor T Cell (CD19 CAR T) Therapy, in Participants With Treatment Refractory Progressive Multiple Sclerosis
Brief Title: A Study of KYV-101, a CD19 CAR T Cell Therapy, in Participants With Treatment Refractory Progressive Multiple Sclerosis
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bruce Cree (Other)
Collaborators: Kyverna Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Bruce Cree, MD, PhD, MAS, Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23-40657
Record Dates: First submitted 2024-06-03; First posted 2024-06-11 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Progressive Multiple Sclerosis
Keywords: multiple sclerosis; CAR-T; University of California, San Francisco (UCSF); progressive multiple sclerosis; treatment refractory progressive multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis | interventions — Biological Products; Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dosing Cohort #1: KYV-101 CAR+ T -- 0.33 ×10^8 cells (Experimental): Five participants will be enrolled at the lower dose (0.33 ×10^8 cells). Once safety and tolerability are adequately assessed, treatment will proceed to the higher dose level.
  Interventions: Biological: KYV-101 (Biological) - 0.33 ×10^8 cells; Drug: Chemotherapy: cyclophosphamide (CYC); Drug: Chemotherapy: fludarabine (FLU)
- Dosing Cohort #2: KYV-101 CAR+ T -- 1×10^8 cells (Experimental): An additional five participants are planned for enrollment at the higher dose level (1×10^8 cells).
  Interventions: Biological: KYV-101 (Biological) - 1 ×10^8 cells; Drug: Chemotherapy: cyclophosphamide (CYC); Drug: Chemotherapy: fludarabine (FLU)

INTERVENTIONS:
Biological: KYV-101 (Biological) - 0.33 ×10^8 cells — KYV-101 is a type of treatment called CAR T-cell therapy. It uses cells from your own immune system, called T-cells, to attack cells that cause inflammation. T-cells are a type of white blood cell.
  Other Names: CAR T-cell therapy
  Arms: Dosing Cohort #1: KYV-101 CAR+ T -- 0.33 ×10^8 cells
Biological: KYV-101 (Biological) - 1 ×10^8 cells — KYV-101 is a type of treatment called CAR T-cell therapy. It uses cells from your own immune system, called T-cells, to attack cells that cause inflammation. T-cells are a type of white blood cell.
  Other Names: CAR T-cell therapy
  Arms: Dosing Cohort #2: KYV-101 CAR+ T -- 1×10^8 cells
Drug: Chemotherapy: cyclophosphamide (CYC) — Participants will receive one 3-day cycle of lymphodepletion with CYC 300 mg/m2 prior to administration of KYV-101.
Drug: Chemotherapy: fludarabine (FLU) — Participants will receive one 3-day cycle of lymphodepletion with FLU 30 mg/m2 prior to administration of KYV-101.

SUMMARY:
The goal of this study is to test a drug called KYV-101 in people who have progressive multiple sclerosis (MS) and who have not responded to standard therapies to slow disease progression. The main questions it aims to answer are:

* What is the highest therapy dose that can be given without causing harm?
* Can this therapy enter the central nervous system?

Participants will be asked to:

* Attend 14 visits plus an 8-day inpatient hospital stay over the course of 58 weeks.
* Complete apheresis and chemotherapy treatments in preparation for KVY-101 therapy.
* Undergo medical and research testing such as physical and neurological exams, MRI, lumbar puncture, blood draws, questionnaires, and vision assessments.

DETAILED DESCRIPTION:
This study will treat up to 10 participants. The primary objective is to characterize central nervous system (CNS) penetration of KYV-101 and its effectiveness of target engagement via elimination of oligoclonal bands (OCB) and/or normalization of immunoglobulin G (IgG) IgG index and to characterize a preliminary safety profile of KYV-101 in treatment-refractory MS.

Pharmacodynamics (PD)/Pharmacokinetics (PK) Objectives

* To characterize the PK and PD of KYV 101 in blood.
* To evaluate changes in PD and disease-related biomarkers.
* To assess the immunophenotype of Chimeric Antigen Receptor (CAR) T cells.

Pharmacodynamics/Pharmacokinetics Endpoints

* CAR-positive T cell counts, CAR transgene level, B-cell counts over time, systemic cytokine concentrations.
* Immunophenotype B and T cells through flow cytometry (including non-CAR T cell and B-cell subsets, if detectable), serum proteins and gene expression analysis.
* CAR T cell phenotypic composition as defined by markers of activation, proliferation, differentiation, and exhaustion (prior to and post infusion).

Abbreviations: CAR=chimeric antigen receptor; PD=pharmacodynamics; PK=pharmacokinetics

Safety/Adverse Event Objectives

* To evaluate for disease re-activation.
* To evaluate the immunogenicity (humoral response) of KYV-101.
* To evaluate the immunogenicity (cellular response) of KYV-101.
* To determine whether RCL is present in participants who receive KYV-101.
* To evaluate changes in long-term humoral response after KYV-101.
* To assess mood patient-reported outcomes (PROs) after infusion of KYV-101.

Safety/Adverse Event Endpoints

* Disease reactivation as defined by the presence of new T2 hyperintense or gadolinium (GAD) enhancing lesions on MRI brain at 8 weeks post-infusion of KYV-101.
* Incidence of detectable anti-KYV-101 antibodies in peripheral blood.
* Incidence of detectable T cells specific to KYV-101 drug product in peripheral blood.
* Detectable replication competent lentivirus (RCL) as measured by surrogate assay (VSV-G qPCR).
* Persistence of IgG antibody titers to common vaccine-related antigens (varicella, measles, mumps, rubella, tetanus).
* Change from baseline in depression/anxiety including Columbia Suicide Severity Rating Scale (C-SSRS).

Abbreviations: RCL=replication competent lentivirus; VSV-G qPCR=vesicular stomatitis virus G glycoprotein quantitative polymerase chain reaction; PRO=patient reported outcomes; C-SSRS=Columbia Suicide severity rating scale

The safety and tolerability of KYV-101 will be evaluated by reported adverse events (AEs), physical examination findings, vital sign measurements, neurological assessment, and laboratory analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must sign a written informed consent form (ICF) prior to any screening procedures.
2. Participant must be 25-70 years of age (inclusive).
3. Clinical diagnosis of MS with evidence of primary or secondary progressive MS based on 2017 International Panel Criteria (Thompson 2018).
4. Historical documented presence of CSF restricted OCBs or elevated IgG Index (reconfirmed on screening).
5. Expanded disability status score (EDSS) score 3.0-7.0
6. Documented evidence of clinical disability progression within the 2 years prior to inclusion, i.e. a) progression of EDSS during the past two years of at least 1 point sustained for at least 6 months if inclusion EDSS is from 3.5 to 5.5 or at least 0.5 point increase sustained for at least 6 months if inclusion EDSS is from 6 to 6.5 or b) increase of Timed Walk 25 (TW25) by at least 20% in the last two years sustained for at least 6 months or c) other well-documented objective worsening despite at least 1 year of prior treatment for progressive forms of MS (including siponimod, and/or anti- B-lymphocyte antigen (CD20) MAb).
7. Adequate organ function as per below:

   Hematology- Hemoglobin > 8 g/dl (without prior red blood cell transfusion within 7 days before the laboratory test) Platelets > 50,000/µL (without transfusion support within 7 days before the laboratory test) Absolute Neutrophil Count (ANC) >1,000/µL (prior growth factor support is permitted but must be without support in the 7 days prior to the laboratory test) Absolute Lymphocyte Count (ALC) > 500/µL IgG > 600 mg/dL Hepatic- Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 1.5 ×upper limit of normal (ULN) Total bilirubin ≤ 1.5 mg/dl, except with Gilbert's syndrome Renal- estimated Glomerular Filtration Rate (eGFR) > 45 mL/min/1.73 m2 (measured by Chronic Kidney Disease (CKD) - Epidemiology Collaboration (EPI) 2021 equation)
8. Positive varicella zoster virus titer. Participants who test seronegative for varicella zoster virus IgG antibodies will be recommended to obtain vaccination prior to Investigational Product (IP) infusion.
9. Participants are recommended to be up to date on other recommended vaccinations, including against Coronavirus Disease (COVID-19)/ Severe Acute Respiratory Syndrome (SARS) Coronavirus 2 (CoV-2), per Centers for Disease Control and Prevention or institutional guidelines for immune-compromised individuals.
10. Women of childbearing potential must have a negative pregnancy test at screening, prior to apheresis, and prior to lymphodepletion chemotherapy using a highly sensitive serum pregnancy test (β- human Chorionic Gonadotropin (hCG)). A woman of childbearing potential is defined as a sexually mature woman who has not undergone a hysterectomy or tubal ligation or who has not been naturally postmenopausal for at least 24 consecutive months.
11. Female participants of childbearing potential who have a fertile male sexual partner must agree to use a highly effective method of contraception (failure rate of < 1% per year when used consistently and correctly) from the time of signing the ICF until 24 months after the KYV-101 infusion. Examples of highly effective method of contraception include:

    * Established use of hormonal methods of contraception associated with inhibition of ovulation (e.g. oral, inserted, injected, implanted, transdermal), provided the participant or male participant's female partner plans to remain on the same treatment throughout the entire study and has been using that hormonal contraceptive for adequate time to ensure effectiveness.
    * Correctly placed copper containing- intrauterine device or intrauterine hormone-replacing system.
    * Female sterilization (bilateral tubal ligation/bilateral salpingectomy or bilateral tubal occlusive procedure (with confirmed occlusion).
    * Sexual abstinence, defined as completely and persistently refraining from all heterosexual intercourse (including during the entire period of risk associated with the study treatments) may obviate the need for contraception only if this is the preferred and usual lifestyle of the participant.
12. Male participants, if not surgically sterilized, must agree to use a highly effective method of contraception until 12 months post IP infusion.
13. Women and men must agree not to donate eggs (ova, oocytes) or sperm, respectively, until at least 12 months after receiving a KYV-101 infusion.
14. Ability to obtain adequate vascular access for leukapheresis procedure (either peripheral line or surgically placed line).

Exclusion Criteria:

1. MS clinical stability on Disease Modifying Therapy (DMT) therapy.
2. Clinical relapse in the two years prior to study entry.
3. Disease other than MS to explain the first demyelinating event; including Aquaporin-4 (AQP4) IgG or Myelin oligodendrocyte glycoprotein (MOG)-IgG seropositivity.
4. Unwilling or unsafe to proceed with cerebral spinal fluid (CSF) exams based on coagulopathy or anatomy or other considerations in the judgment of the study investigator.
5. Unwilling or unsafe to proceed with MRI.
6. History of allogeneic or autologous stem cell transplant or solid organ transplant.
7. Prior treatment CAR-T or gene therapy product directed at any target.
8. Prior treatment with mitoxantrone, cladribine or alemtuzumab.
9. Need for ongoing anticoagulation.
10. Presence of hypogammaglobulinemia defined as IgG < 600 mg/dL.
11. Plan to receive live, attenuated vaccine after signing ICF (inactive vaccines, like the influenza vaccine, are allowed).
12. Unable to interrupt autoimmune disease therapy prior to apheresis
13. Serologic status reflecting active hepatitis B or C infection. Patients who are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment. (PCR positive patients will be excluded.) Patients who are positive for hepatitis B core antibody will be required to remain on appropriate prophylactic antiviral therapy (e.g. with entecavir) for the duration of the study.
14. Positive serology for human immunodeficiency virus (HIV).
15. History of progressive multifocal leukoencephalopathy.
16. Untreated active or untreated latent tuberculosis or documented completed treatment without a negative chest X-ray (CXR) that shows no evidence of active Tuberculosis (TB).
17. Primary immunodeficiency as defined by a known genetic disorder.
18. History of splenectomy.
19. Impaired cardiac function or clinically significant cardiac disease including:

    1. Unstable angina or myocardial infarction or coronary artery bypass graft (CABG) within 6 months prior to apheresis.
    2. New York Heart Association (NYHA) stage III or IV congestive heart failure.
    3. History of clinically significant cardiac arrhythmia (eg, ventricular tachycardia), complete left bundle branch block, high-grade atrioventricular (AV) block, or QT prolongation.
    4. Inadequate cardiac function defined as left ventricular ejection fraction (LVEF) < 40% as assessed by echocardiogram within 3 months of screening. Repeat testing may occur at Investigator's discretion.
20. Previous or concurrent malignancy with the following exceptions:

    1. Adequately treated basal cell or squamous cell carcinoma (adequate wound healing is required prior to screening).
    2. In situ carcinoma of the cervix or breast, treated curatively and without evidence of recurrence for at least 3 years prior to screening.
    3. A primary malignancy which has been completely resected, or treated, and is in complete remission for at least 5 years prior to screening.
21. Serious and/or uncontrolled medical condition that, in the investigator's judgment, would cause unacceptable safety risk, interfere with study procedures or results, or compromise compliance with the protocol, such as:

    1. Active, uncontrolled, viral, bacterial, or systemic fungal infection.
    2. Chronic viral, bacterial, or systemic fungal infection that may be reactivated during treatment.
    3. Requirement of supplemental oxygen to maintain oxygen saturation.
    4. Clinical evidence of dementia.
    5. A thromboembolic event within 6 months prior to apheresis.
    6. On anti-coagulation agents that would be unsafe to transiently hold for medical procedures.
    7. Uncontrolled Diabetes Mellitus (DM) or Hypertension (HTN).
22. Major surgery within 4 weeks prior to apheresis or planned within 4 weeks after KYV-101 administration. For surgery planned after 4 weeks post KYV-101 administration, discuss with the investigator.
23. History of any other neurologic disorder or medical condition the investigator considers would increase the risk for the participant, including seizure disorders.
24. Contraindications or life-threatening allergies, hypersensitivity, or intolerance to KYV-101 or its excipients, including dimethyl sulfoxide; cyclophosphamide (CYC) or fludarabine (FLU); or tocilizumab.
25. Pregnant or breastfeeding; or plans to become pregnant or breastfeed within 24 months after receiving the KYV-101 infusion.
26. Unwilling to participate in long-term follow up for safety monitoring after CAR-T therapy.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
The presence of CAR-T cells in CSF following their peak expansion in peripheral blood. | Screening to Week 48
  To surmise CNS penetration of CAR-T cells.
The incidence and severity of adverse events and dose-limiting toxicities. | Screening to Week 48
  * Disease reactivation as defined by the presence of new T2 hyperintense or GAD enhancing lesions on MRI brain at 8 weeks post-infusion of KYV-101.
  * Incidence of detectable anti-KYV-101 antibodies in peripheral blood.
  * Incidence of detectable T cells specific to KYV-101 drug product in peripheral blood.
  * Detectable replication competent lentivirus as measured by surrogate assay (VSV-G qPCR).
  * Persistence of IgG antibody titers to common vaccine related antigens (varicella, measles, mumps, rubella, tetanus).
  * Change from baseline in depression/anxiety including C-SSRS.

SECONDARY OUTCOMES:
The proportion of participants in whom reduction of CSF OCB and/or normalization of CSF IgG Index are detected. | Screening to Week 48
  To characterize the evidence of target engagement within the CNS of KYV-101.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Cree, MD, PhD, MAS, Principal Investigator — University of California, San Francisco; Sasha Gupta, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, Multiple Sclerosis Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No